CLINICAL TRIAL: NCT06837701
Title: The True Face of the Pyramid; Physical Activity Level and Cardiovascular Risk in Patients With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ebru Calik Kutukcu, Professor, Hacettepe University
Other Study IDs: SBA 24/664
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Cardiovascular Disease; Physical Activity
Keywords: breast cancer; Cardiovascular disease; Physical activity
MeSH Terms: conditions — Breast Neoplasms; Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of morbidity and mortality worldwide. Many risk factors are thought to be important in the development of CVD; however, some risk factors can be controlled. Regular physical activity (PA) is recommended for the entire population for the primary prevention of CVD. PA and physical health are also believed to reduce other CVD risk factors such as body mass index, blood pressure and stress. Although oncological outcome is the most important factor for breast cancer survivors, CVD has emerged as an important cause of death among them. In particular, CVD mortality is known to increase 7 years after breast cancer diagnosis, and death due to CVD is more common in older patients than death from cancer. Higher levels of physical activity compared to low levels measured prior to breast cancer diagnosis were associated with statistically significantly lower all-cause mortality among women diagnosed with breast cancer. For breast cancer survivors, increasing PA during and after treatment has been reported to be safe and effective in improving cancer survival, alleviating cancer-related symptoms and improving quality of life. However, there is a lack of evidence regarding the effect of PA on cardiovascular outcomes in long-term breast cancer survivors.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of morbidity and mortality worldwide. Many risk factors are thought to be important in the development of CVD; however, some risk factors can be controlled. Regular physical activity (PA) is recommended for the entire population for the primary prevention of CVD. PA and physical health are also believed to reduce other CVD risk factors such as body mass index, blood pressure and stress. Although oncological outcome is the most important factor for breast cancer survivors, CVD has emerged as an important cause of death among them. In particular, CVD mortality is known to increase 7 years after breast cancer diagnosis, and death due to CVD is more common in older patients than death from cancer. Higher levels of physical activity compared to low levels measured prior to breast cancer diagnosis were associated with statistically significantly lower all-cause mortality among women diagnosed with breast cancer. For breast cancer survivors, increasing PA during and after treatment has been reported to be safe and effective in improving cancer survival, alleviating cancer-related symptoms and improving quality of life. However, there is a lack of evidence regarding the effect of PA on cardiovascular outcomes in long-term breast cancer survivors.

This study aims to investigate the determination of optimal walking or moderate to vigorous PA in patients categorised according to their cardiovascular health status. We also aimed to evaluate the association of different levels of physical activity with cardiovascular risk in different age groups after breast cancer.

Demographic information: Participants' age, diagnosis, medical history (time since surgery (months), type of lymphedema, treatments received for lymphedema, radiotherapy (number of days), chemotherapy (number of cycles), type of surgery (lumpectomy, segmental mastectomy, modified radical mastectomy, radical mastectomy), occupation, body weight (kg), height (cm), body mass index (kg/m2), lean muscle mass and fat percentage will be assessed as part of anthropometric evaluation (Tanita Inner Scan BC 532, Tokyo, Japan). Waist and hip circumference measurements will be recorded. BMI, dominant and affected side, medical history, family history, lifestyle characteristics (smoking, exercise habits, alcohol intake), monthly income level will be recorded.

Assessment of Physical Activity Level: Physical activity level will be assessed with a triaxial accelerometer. SenseWear Armband (SWA) (Armband Model MF-SW, BodyMedia, Pittsburgh, USA) metabolic holter device with triaxial accelerometer sensors that detect skin temperature, galvanic skin response, heat flow, movement and position will be used to objectively measure activity level and energy consumption. After the configuration of the device is made, it will be given to the individuals to be worn for 7 consecutive days or more. Individuals will be asked to remove the device only when taking a shower and in situations requiring contact with water, such as swimming, and then dry the arm and reinsert the device. The device will be worn as described in the manual, with the left arm over the triceps muscle, making sure that the sensors are in contact with the person's arm, and adjusting the band tightness according to the person's arm. Individuals will be asked to continue their daily life activities as usual while wearing the device. The data obtained from the device will be recorded together with the individuals' date of birth, height, body weight, gender, dominant hand and smoking status.

Total energy expenditure, active energy expenditure, average number of steps, average MET, average physical activity index (PAL), average distance, duration of physical activity, duration of mild physical activity (<1.5 MET), duration of moderate physical activity (3-6 MET), duration of vigorous physical activity (6-9 MET), duration of very vigorous physical activity (>9 MET), duration of lying down, average sleep time and sleep efficiency data will be obtained from the device.

Assessment of comorbidity level: It will be assessed with the Charlson Comorbidity Index. This index was developed by Charlson et al. This index was developed by Charlson et al. in a study involving 559 patients in order to predict mortality due to chronic diseases. It is an easily applicable scale that predicts the risk of death due to comorbidities. Diseases associated with 1-year mortality were determined and weight scores were determined according to risk status. This measure was then applied on 686 patients and shown to be a good predictor of survival. It is scored between 0-6 according to comorbidities. As the total score increases, the risk of mortality increases. Especially a score of 3 and above increases the risk of mortality.

Quality of life assessment: The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30), which was developed specifically for cancer patients, will be used to assess the quality of life of the patients in the study.When calculating the functional status score, a raw score (HP) is first calculated by taking the arithmetic mean of the answers given to the relevant 15 questions. Since the highest score is '4' and the lowest score is '1', the difference between them gives the interval value of '3'. Functional status=(1-(HP-1)\/interval)×100 When calculating the functional status sub-headings, the same formula is used by taking the arithmetic mean of the relevant questions. When calculating the symptom score, HP is first calculated by taking the arithmetic mean of the answers given to the relevant 13 questions. Since the highest score is '4' and the lowest score is '1', the difference between them gives the interval value of '3'. Symptom Score= ((HP-1)\/interval)×100 When calculating the subheadings of the symptom section, the same formula is used by taking the arithmetic averages of the relevant questions. When calculating the general health status score, the HP is calculated by taking the arithmetic mean of the answers given to the relevant 2 questions.Since the highest score is '7' and the lowest score is '1', the difference between these two questions gives a range value of '6'. General health status score=((HP-1)/interval)×100 The questionnaire was adapted into Turkish by Güzelant et al. and its validity and reliability were determined for the Turkish population.

Cardiovascular Disease Risk Scoring: SCORE2. The SCORE risk scoring was developed by analysing data from studies in 12 European countries, with more than 200,000 participants, approximately 3 million annual follow-ups and more than 7,000 cardiovascular deaths. In the SCORE table, which has a high applicability in primary care, 10-year CVD event risk is determined using age, gender, total cholesterol, smoking status and blood pressure values. All atherosclerotic deaths (not only deaths due to CAD) are taken into account in the risk calculation and stroke-related deaths can be separated from CAD-related deaths when desired. Studies in the SCORE database have shown that HDL-cholesterol may have a significant effect on risk calculation. When HDL-cholesterol values are included, SCORE tables show that the risk changes at all risk levels, at all ages and sexes. The updated SCORE algorithm, SCORE2, incorporates the effect of the non-HDL-cholesterol value and estimates an individual's 10-year risk of fatal and non-fatal CVD events (myocardial infarction, stroke) in apparently healthy people aged 40-69 years with risk factors. SCORE2 and SCORE2-OP are calibrated according to four country clusters (low, intermediate, high and very high CVD risk) grouped according to national CVD mortality rates published by WHO. Turkey is in the high-risk countries group. The risk calculated according to the SCORE system is considered low risk if <1%, medium risk if 1-4%, high risk if 5-9%, and very high risk if 10% and above. According to the SCORE2 system, those under the age of 50 are considered to be at low-moderate risk if <2.5%, high risk if 2.5%-7.5%, and very high risk if 7.5% and above. In those over 50 years of age, <5% is considered low-moderate risk, 5-10% is considered high risk, and 10% and above is considered very high risk.

Cardiovascular Diseases Risk Factors Knowledge Level Scale (CARRIF-BD): It was developed by Arıkan et al. in 2009 and validity and reliability studies were conducted. While the first four items of the scale consisting of twenty-eight items are related to the characteristics of cardiovascular disease, preventability and age factor, 15 items question the risk factors and nine items question the result of change in risk behaviours. The items in the scale are presented to the participants in the form of a complete sentence that can be true or false and the participants are asked to answer these statements as "Yes", "No" or "I don't know". In the scale, 1 point is given for each correct answer and 6 questions are scored in the opposite direction. Scores between 0-28 can be obtained from the scale. The higher the score, the higher the level of knowledge. Arıkan et al. found the Cronbach alpha value of the scale as 0.76. However, it was stated that the scale was suitable for determining the cardiovascular disease risk knowledge of all individuals in Turkey.

Hospital Anxiety and Depression Scale (HAD): The HAD is a four-point Likert-type scale developed by Zigmond and Snaith to determine the risk of anxiety and depression in patients and to measure the level and severity change. It contains a total of 14 questions and odd numbers measure anxiety and even numbers measure depression. The Turkish validity and reliability of the form was performed by Aydemir and it was determined that the scale was safe in terms of screening depression and anxiety symptoms in patients with physical illness. It has anxiety (HAD-A) and depression (HAD-D) subscales. As a result of the study conducted in Turkey, a cut-off score of 10/11 was found for the anxiety subscale and 7/8 for the depression subscale. Accordingly, those above these scores are considered to be at risk. The scoring of each item in the scale is different. Items 1, 3, 5, 6, 8, 10, 11 and 13 show gradually decreasing severity and the scoring is 3, 2, 1, 0. On the other hand, items 2, 4, 7, 9, 12 and 14 are scored as 0, 1, 2, 3. For the anxiety subscale, the scores of items 1, 3, 5, 7, 9, 11 and 13 are summed; for the depression subscale, the scores of items 2, 4, 6, 8, 10, 12 and 14 are summed. The lowest score that patients can get from both subscales is 0 and the highest score is 21.

Type D Personality Scale (DS-14): Type D Scale-14 (DS-14) was developed to assess negative affectivity (NA), social inhibition (SI) and type D personality. The DS-14 consists of a total of 14 items and two subscales measuring NA and SI. Each item is a Likert-type scale scored between 0-4. The cut-off point of both subscales is ≥10 (28). Both subscales have good test-retest validity and high internal validity.

Assessment of functional exercise capacity: Functional exercise capacity will be assessed with 6DYT, a submaximal exercise test. The standard protocol is to be performed in a 30-metre straight corridor. The participant, wearing comfortable clothing and shoes, is given standard instructions during the test and is asked to walk as fast as he/she can walk for 6 minutes. Heart rate (HR) and oxygen saturation (SpO2) values will be recorded before, after and during the test with a wristband worn on the hand and a portable field testing system pulse oximeter attached to the finger at the end. Dyspnoea, leg and body fatigue perceptions will be evaluated with the Modified Borg Scale (MBS) between 0-10 points.

ELIGIBILITY:
Inclusion Criteria:

1. To be between the ages of 40-80 years,
2. Volunteering to participate in the research,
3. At least 15 months after breast cancer surgery,
4. 6 months after active breast cancer treatment (ie surgery/chemotherapy)
5. Having no problem in reading and/or understanding the scales and being able to cooperate with the tests.

Exclusion Criteria:

1. Presence of active infection,
2. Having a neurological disease or other clinical diagnosis that may affect cognitive status,
3. Having musculoskeletal and neurological disease, symptomatic heart disease, previous lung surgery and malignant disease that may affect exercise performance.
4. Presence of unstable hypertension or diabetes mellitus

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Population:
  Patients between the ages of 40-80 years who were diagnosed with breast cancer in Hacettepe University Hospital, Department of Internal Medicine, Department of Medical Oncology and volunteered to participate in the study will be included in the study.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Physical Activity Level | One Year
  Physical activity level was assessed using a multisensorial PA monitor. The SenseWear Armband (Armband Model MF-SW, BodyMedia, Pittsburgh, USA) was worn on the back of the left-side upper arm over the triceps for at least 7 consecutive days, except for times requiring contact with water, such as bathing and swimming. The monitor estimates energy expenditure using measurements from tri-axial accelerometers and sensors (galvanic skin response, heat flux, and skin temperature). The measured outputs of the SWA is step count
Cardiovascular Disease Risk Scoring | One Year
  SCORE2
Functional exercise capacity | one year
  6 minutes walk test

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Calik Kutukcu, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, State, Turkey (Türkiye)